CLINICAL TRIAL: NCT03337334
Title: Effects of High Amplitude and Focused tACS on Entraining Physiological Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Ahmad Khatoun, Principal Investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: S57869
Record Dates: First submitted 2017-11-01; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Tremor, Limb
MeSH Terms: conditions — Tremor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Focused stimulation (Other): Stimulation frequency is set similar to that of the tremor and the amplitude is set up to 2 mA peak amplitude (reduced if not uncomfortable). One 5*5 cm2 square patch electrodes are placed over the Motor cortex and the Prefrontal cortex respectively and a common return electrode of 10*10 cm2 over the ankle. Each subject follows three sessions of 12 min length each. During each session the tremor is measured while interleaving between Motor cortex stimulation, Prefrontal cortex stimulation and No stimulation. By the end of each session we get 4 min of Motor Cortex stimulation, 4 min of Prefrontal Cortex stimulation and 4 min of No stimulation.
  Interventions: Device: tACS at tremor frequency
- Focused stimulation (Other): Stimulation frequency is set similar to that of the tremor and the amplitude is set up to 5 mA peak amplitude (with the help of local anesthetic cream and amplitude is reduced if not uncomfortable). A set of 4*1 gel-filled cup-electrodes is placed over each of motor cortex and the occipital cortex respectively. Each subject follows three sessions of 12 min length each. During each session the tremor is measured while interleaving between Motor cortex stimulation, Occipital cortex stimulation and No stimulation. By the end of each session we get 3 min of Motor Cortex stimulation, 3 min of occipital Cortex stimulation and 6 min of No stimulation.
  Interventions: Device: tACS at tremor frequency

INTERVENTIONS:
Device: tACS at tremor frequency — tACS applied between the stimulation electrodes at tremor frequency

SUMMARY:
Transcranial alternating current stimulation (tACS) is a noninvasive neuromodulation method that works by passing alternating electric current between electrodes where at least one of them is attached to the head. While tACS applied over the motor cortex at the general applied amplitude (1 mA) and using patch electrodes has been shown to entrain physiological tremor in healthy volunteers, the aim of this study is to test the feasibility of using high-amplitude tACS and to assess the effect of different electrode montages and stimulation sites in entraining physiological tremor. First, 10 subjects (arm 1) will be stimulated with 2 mA current amplitude applied between saline soaked patch square electrodes and comparison will be done between motor cortex stimulation and peripheral cortex stimulation. Then, 10 subjects (arm 2) will be stimulated using focused 4x1 montage with gel-filled cup-electrodes and 5 mA amplitude and comparison will be made between motor cortex and occipital cortex stimulation. Three outcome measurements will be measured during the experiments which are: tremor entrainment, phosphene intensity and phosphene threshold.

ELIGIBILITY:
Inclusion Criteria:

* Above 18
* signed informed written consent

Exclusion Criteria:

* Pregnancy
* History of Epilepsy
* Family history of Epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Tremor-stimulation phase entrainment | During the 36 minutes of all sessions (3 sessions each of is 12 minutes)
  phase locking value was calculated between the tremor signal measured using accelerometer and the stimulation signal

SECONDARY OUTCOMES:
Phosphene rating | Measured up to 5 minutes before the start of the stimulation sessions and lasts for 10 seconds of stimulation after which the subject gives the rating
  The subject is asked to rate the phosphene intensity during the stimulation using a visual analog scale from 0 to 10. Zero means no phosphene is perceived and the number starts to increase as the phosphene perception intensity increases to reach 10 if the subject observe only a white view
Phosphene threshold | Measured 3 minutes before the start of the stimulation sessions and lasts up to 2 minutes. Stimulation at each amplitude lasts for 10 sec.
  Stimulation amplitude at which the subject starts to perceive phosphene. Stimulation starts with 0 mA amplitude and then increased gradually until phosphene is perceived (or reaching maximum amplitude).

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-01): https://cdn.clinicaltrials.gov/large-docs/34/NCT03337334/Prot_SAP_000.pdf